CLINICAL TRIAL: NCT01730183
Title: To Study the Safety and Efficacy of Autologous Bone Marrow Stem Cells in Patients With Spinal Cord Injury (SCI)
Brief Title: To Study the Safety and Efficacy of Autologous Bone Marrow Stem Cells in Patients With Spinal Cord Injury
Acronym: ABSCI
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Max Institute of Neurosciences (Industry)
Responsible Party: Principal Investigator, Yashbir Dewan, Consultant Neurosurgeon, Max Institute of Neurosciences
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TPSC/POC/BMSC/SCI; NCT01490242 (obsolete NCT alias)
Record Dates: First submitted 2012-11-15; First posted 2012-11-21 (Estimated); Last update posted 2012-11-21 (Estimated); Status verified 2012-11

CONDITIONS: Spinal Cord Injury
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Bone marrow derived stem cells (Experimental): Autologous Bone Marrow derived Stem Cells(BMSC) transplanted intrathecally into patients with spinal cord injury.
  Interventions: Other: Bone marrow derived stem cells

INTERVENTIONS:
Other: Bone marrow derived stem cells — Intrathecal administration of autologous bone marrow derived stem cells upto a cell dose of equal or greater than 10(8)BMMNCs.
  Other Names: Bone Marrow derived Mononucleated stem cell (BMMNCs)

SUMMARY:
This is a Phase I/II, multicenter, prospective, non-randomized, open label study to evaluate the safety/efficacy of autologous bone marrow-derived stem cell transplantation in spinal cord injury patients.

DETAILED DESCRIPTION:
Spinal cord injury (SCI) is a traumatic disorder resulting in a functional deficit that usually leads to severe and permanent paralysis and the projected data related to the burden of spinal cord injuries across the globe is quite alarming. Pharmacological and rehabilitation therapies to SCI have got limited effect. There is definitely an urgent need for finding different methods of treatment for these patients who cannot undergo established modalities of treatment or these have been tried unsuccessfully. Another promising therapeutic approach for SCI is "Stem cell transplantation". Bone marrow derived stem cells have been shown to promote anatomical and functional recovery in animal models of SCI by promoting tissue sparing, axonal regeneration, and remyelination. In our present study, we want to evaluate the safety and efficacy of autologous bone marrow derived stem cells surgically transplanted intrathecally into patients with spinal cord injury.

ELIGIBILITY:
Inclusion Criteria:

1. Traumatic injury of the spinal cord (below C5 level) occurring within 6 months to 8 years prior to treatment, resulting in a sustained and complete / Partial loss of sensory and motor function below the injury (ASIA Category A, B and C ).
2. Confirmation spinal cord injury level (Patients with complete or partial transection/damage by MRI).
3. Those provide fully informed consent.
4. The level of spinal cord injury must be below C4.

Exclusion Criteria:

1. Spinal vertebral instability.
2. Major concurrent medical illness (e.g. carcinoma, auto-immune disease,)
3. ASIA Impairment Scale category other than D & E.
4. Lactating and pregnant women.
5. Syringomyelia is also an exclusion criterion but an exemption can be made for a patient with a stable syrinx.
6. Platelet count greater than 100 thousand/µl at screening.
7. Hematocrit less than 30% prior to bone marrow aspiration.
8. Patients with major and current psychiatric illness.
9. Significant traumatic brain injury associated with the spinal cord injury.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 15 (Estimated)
Dates: Start 2012-11; Primary Completion 2014-11 (Estimated); Study Completion 2014-11 (Estimated)

PRIMARY OUTCOMES:
Number of participants with adverse events as a measure of safety and tolerability. | 18 months
  The measure is the number of adverse events following intrathecal administration of autologous bone marrow derived stem cells in spinal cord injury patients.

SECONDARY OUTCOMES:
Significant improvement in the ASIA scores by the assessment motor, sensory and sphincteric function. | 18 months
  * Improvement in the functional Independence as measured by Spinal Cord Independence Measure (SCIM III). [ Time Frame: Baseline and 18 months ] [ Designated as safety issue: No ]
  * Improvement in the pain sensation score as measured by Bryce/Ragnarsson SCI pain taxonomy (BR-SCI-PT). [ Time Frame: Baseline and 18 months ] [ Designated as safety issue: No ]
  * Significant Changes in the muscle tone as indicated by Modified Ashworth Scale (MAS). [ Time Frame: Baseline and 18 months ] [ Designated as safety issue: No ]
  * Improvement in the Clinical Outcome Variable Scale (COVS) score. [ Time Frame: Baseline and 18 months ] [ Designated as safety issue: No ]

CONTACTS AND LOCATIONS:
Overall Officials: Yashbir Dewan, MS, MCh, Principal Investigator — Max Healthcare; Yashbir Dewan, MS, MCh, Study Chair — Max Helathcare
Locations (1):
- Max Super speciality Hospital, Dehradun, Uttrakhand, India

REFERENCES:
- [Background] Geffner LF, Santacruz P, Izurieta M, Flor L, Maldonado B, Auad AH, Montenegro X, Gonzalez R, Silva F. Administration of autologous bone marrow stem cells into spinal cord injury patients via multiple routes is safe and improves their quality of life: comprehensive case studies. Cell Transplant. 2008;17(12):1277-93. doi: 10.3727/096368908787648074. PMID 19364066